CLINICAL TRIAL: NCT01428817
Title: Carbetocin at Elective Cesarean Delivery: A Dose Finding Study (Part 2)
Brief Title: Carbetocin at Elective Cesarean Delivery Part 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Dr. Jose C.A. Carvalho, Mount Sinai Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-02
Record Dates: First submitted 2011-09-01; First posted 2011-09-05 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Postpartum Hemorrhage
Keywords: pregnancy; postpartum hemorrhage; Cesarean delivery; carbetocin
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — carbetocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Carbetocin 20mcg (Active Comparator)
  Interventions: Drug: Carbetocin
- Carbetocin 40mcg (Active Comparator)
  Interventions: Drug: Carbetocin
- Carbetocin 60mcg (Active Comparator)
  Interventions: Drug: Carbetocin
- Carbetocin 80mcg (Active Comparator)
  Interventions: Drug: Carbetocin
- Carbetocin 100mcg (Active Comparator)
  Interventions: Drug: Carbetocin

INTERVENTIONS:
Drug: Carbetocin — 20mcg carbetocin, IV, over 1 minute following delivery of the fetal head.
  Other Names: Duratocin
  Arms: Carbetocin 20mcg
Drug: Carbetocin — 40mcg carbetocin, IV, over 1 minute following delivery of the fetal head.
  Other Names: Duratocin
  Arms: Carbetocin 40mcg
Drug: Carbetocin — 60mcg carbetocin, IV, over 1 minute following delivery of the fetal head.
  Other Names: Duratocin
  Arms: Carbetocin 60mcg
Drug: Carbetocin — 80mcg carbetocin, IV, over 1 minute following delivery of the fetal head.
  Other Names: Duratocin
  Arms: Carbetocin 80mcg
Drug: Carbetocin — 100mcg carbetocin, IV, over 1 minute following delivery of the fetal head.
  Other Names: Duratocin
  Arms: Carbetocin 100mcg

SUMMARY:
Post-partum hemorrhage (PPH) is a major cause of maternal death worldwide. Oxytocin is the most common uterotonic drug used to prevent and treat PPH in North America, however, there are some limitations to its use. Oxytocin has a very short duration of action, which requires a continuous infusion to achieve sustained uterotonic activity. The Society of Obstetricians and Gynecologists of Canada (SOGC) has recently recommended a single 100mcg dose of carbetocin at elective Cesarean delivery to promote uterine contraction and prevent post partum hemorrhage (PPH), in lieu of the more traditional oxytocin regimens. Carbetocin lasts 4 to 7 times longer than oxytocin, with a similar side effect profile and apparent greater efficacy rate. However, a dose response to determine the minimum effective dose of carbetocin has not yet been published. The investigators hypothesize that the minimum effective dose (ED90) is above 20mcgs and below 80mcgs in women undergoing elective Cesarean delivery.

DETAILED DESCRIPTION:
The Society of Obstetricians and Gynecologists of Canada (SOGC) recently recommended a 100mcg intravenous bolus dose of carbetocin following Cesarean delivery.

Studies thus far show that carbetocin may be just as effective as oxytocin in promoting uterine contraction, with a similar side effect profile. In addition, patients receiving carbetocin may experience less blood loss, and require less additional uterotonics when compared with oxytocin. A dose response study conducted by Cordovani et al suggested no difference in efficacy of uterine contraction for doses of carbetocin between 80-120mcg. Additionally, hypotension was noted for all dose groups studied.

The results of this follow-up study will define the minimum required dose of carbetocin for uterine contraction, thus minimizing unnecessary side effects, improving quality and safety of patient care. It may also contribute in establishing carbetocin as a substitute to oxytocin for elective cesarean section at our institution as well as others.

ELIGIBILITY:
Inclusion Criteria:

* All patients planned for elective cesarean delivery under spinal anesthesia.
* All patients who give written informed consent to participate in this study.

Exclusion Criteria:

* All patients who refuse to give written informed consent.
* All patients who claim allergy or hypersensitivity to carbetocin or oxytocin.
* All patients with conditions that predispose to uterine atony and postpartum hemorrhage such as placenta previa, multiple gestation, preeclampsia, eclampsia, macrosomia, polyhydramnios, uterine fibroids, previous history of uterine atony and postpartum bleeding, or bleeding diathesis.
* All patients with hepatic, renal, and vascular disease,
* All patients requiring general anesthesia prior to the administration of the study drug.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2011-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Uterine tone | 2 minutes
  The obstetrician will assess uterine tone by palpation. Uterine tone will be rated as satisfactory (firm) or unsatisfactory (boggy).

SECONDARY OUTCOMES:
Uterine tone | 2 hours
  Uterine tone will be assessed by palpation 2 hours post-delivery by the nurse/obstetrician in the recovery room.
Blood loss | 48 hours
  Blood loss will be calculated through the difference in hematocrit values assessed prior to and at the end of 48 hours after the cesarean section.
Side effects | 2 hours
  Any of the following will be noted up to 2 hours post delivery: systolic blood pressure < 80% of pre-delivery values, tachycardia > 30% pre-delivery levels, bradycardia < 30% pre-delivery levels, other dysrhythmias, nausea, vomiting, chest pain, shortness of breath, headache, flushing, others

CONTACTS AND LOCATIONS:
Overall Officials: Jose CA Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Anandakrishnan S, Balki M, Farine D, Seaward G, Carvalho JC. Carbetocin at elective Cesarean delivery: a randomized controlled trial to determine the effective dose, part 2. Can J Anaesth. 2013 Nov;60(11):1054-60. doi: 10.1007/s12630-013-0028-2. Epub 2013 Sep 25. PMID 24158878